CLINICAL TRIAL: NCT02531022
Title: A Randomized, Controlled Trial Evaluating Methods to Use Physical Activity to Improve Outcomes After Acute Coronary Syndrome
Brief Title: Evaluating Increasing Physical Activity After Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 823025
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Physical Activity; Acute Coronary Syndrome
MeSH Terms: conditions — Motor Activity; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Participants will be given standard exercise recommendations that are given to all patients based on the federal guidelines. They will monitor their step counts using a wearable device and receive daily feedback.
  Interventions: Behavioral: Daily feedback
- Intervention (Experimental): Participants will be given a wearable device to monitor daily step counts with automated daily feedback on goal attainment via text message or email. A baseline step count will be calculated for each participant (weeks 1-2) and then they will be given a daily step goal with an increase of 15 percentage point each week during the 8-week ramp-up period (weeks 3-10) with a maximum goal of 10,000 steps. Then they'll be asked to maintain that step count (maintenance period). During the ramp-up and maintenance period they'll have a financial incentive of $14 allocated each week and $2 taken away each day the goal is not achieved. They'll be followed up for 8 weeks without incentives
  Interventions: Behavioral: Financial incentive; Behavioral: Daily feedback

INTERVENTIONS:
Behavioral: Financial incentive — A daily financial incentive framed as a loss of $2 each day goal is not acheived
  Arms: Intervention
Behavioral: Daily feedback — Daily feedback from an activity tracking device worn on the wrist to track step counts and sleep patterns

SUMMARY:
This study will use a randomized, controlled trial to test the effectiveness of a home-based physical activity program using wearable devices and financial incentives. All participants in will establish a baseline step count during the first two weeks and then proceed to a 16-week intervention period and 8-week follow-up period.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of mortality in the United States. Among patients that survive an acute myocardial infarction (AMI), cardiac rehabilitation (CR) has been demonstrated to effectively reduce risk of re-infarction, cardiac mortality, and all-cause mortality. However, despite cardiac rehabilitation being a Class I (standard of care) recommendation in multiple American Heart Association acute myocardial infarction guidelines, more than 80% of eligible patients do not receive appropriate cardiac rehabilitation and much of this is due to challenges in access to these programs. Recent innovations in technology allow us to passively monitor an individual's physical activity using wearable devices. Incentives designed using insights from behavioral economics have been demonstrated to motivate device engagement and behavior change. A remotely-monitored cardiac rehabilitation program could improve access for many individuals and potentially be more cost-effective because it is less resource- and personnel-intensive. The objective of this study is to use a randomized, controlled trial to test the effectiveness of a home-based physical activity program using wearable devices and financial incentives.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. ability to read and provide informed consent to participate in the study;
3. History of a) acute coronary syndrome (unstable angina, non-ST segment elevation myocardial infarction or ST segment elevation myocardial infarction); or b) patients having undergone coronary catheterization for suspected coronary artery disease.

Exclusion Criteria:

1. Inability to provide informed consent;
2. does not have daily access to a smartphone compatible with the wearable device;
3. unable or unwilling to complete the baseline 6-minute walk test and return to perform the 6-minute walk test at 10 and 18 weeks;
4. already enrolled in an exercise cardiac rehabilitation program prior to hospital admission;
5. hemodynamic instability or New York Heart Association III-IV heart failure;
6. any other medical conditions that would prohibit participation in an 18-week physical activity program;
7. not being discharged to home if recently admitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortunato M, Adusumalli S, Chokshi N, Harrison J, Rareshide C, Patel M. Usability of Wearable Devices to Remotely Monitor Sleep Patterns Among Patients With Ischemic Heart Disease: Observational Study. JMIR Form Res. 2020 Apr 7;4(4):e14508. doi: 10.2196/14508. PMID 32254044
- [Derived] Chokshi NP, Adusumalli S, Small DS, Morris A, Feingold J, Ha YP, Lynch MD, Rareshide CAL, Hilbert V, Patel MS. Loss-Framed Financial Incentives and Personalized Goal-Setting to Increase Physical Activity Among Ischemic Heart Disease Patients Using Wearable Devices: The ACTIVE REWARD Randomized Trial. J Am Heart Assoc. 2018 Jun 13;7(12):e009173. doi: 10.1161/JAHA.118.009173. PMID 29899015

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Exercise/Control: Participants were given standard exercise recommendations that are given to all patients based on the federal guidelines. They also monitored their step counts using a wearable device and received daily feedback.
- Daily Feedback With Financial Incentive: Participants were given standard exercise recommendations that are given to all patients based on the federal guidelines. They also monitored their step counts using a wearable device, received daily feedback and were eligible for a financial incentive if their goals were achieved.
  Daily feedback: Daily feedback from an activity tracking device worn on the wrist to track step counts and sleep patterns Financial incentive: A daily financial incentive framed as a loss of $2 each day goal is not achieved
Period: Overall Study
Arm/Group | Standard Exercise/Control | Daily Feedback With Financial Incentive
Started | 55 | 50
Completed | 55 | 48
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control: Participants were given standard exercise recommendations that are given to all patients based on the federal guidelines. They also monitored their step counts using a wearable device and received daily feedback.
- Intervention: Participants were given standard exercise recommendations that are given to all patients based on the federal guidelines. They also monitored their step counts using a wearable device, received daily feedback and were eligible for a financial incentive if their goals were achieved.
  Daily feedback: Daily feedback from an activity tracking device worn on the wrist to track step counts and sleep patterns Financial incentive: A daily financial incentive framed as a loss of $2 each day goal is not achieved
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 55 | 50 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.5) | 60 (9.5) | 59.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 37 | 36 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 38 | 38 | 76
  Black non-Hispanic | 14 | 8 | 22
  Other | 3 | 4 | 7
Education [Count of Participants; unit: Participants]
  Some high school | 3 | 3 | 6
  High school graduate | 10 | 12 | 22
  Some college or specialized training | 18 | 8 | 26
  College graduate | 24 | 26 | 50
  Missing | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants]
  Single | 11 | 12 | 23
  Married | 35 | 29 | 64
  Other | 9 | 9 | 18
Insurance [Count of Participants; unit: Participants]
  Private | 28 | 24 | 52
  Medicare | 24 | 21 | 45
  Medicaid | 2 | 4 | 6
  Military | 1 | 1 | 2
Annual household income [Count of Participants; unit: Participants]
  Less than $50,000 | 21 | 18 | 39
  $50,000 to $100,000 | 17 | 7 | 24
  Greater than $100,000 | 12 | 17 | 29
  Missing | 5 | 8 | 13
Baseline step count [Mean (Standard Deviation); unit: steps] | 6577 (3084) | 7205 (3246) | 6876 (3163)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (5.6) | 31.0 (6.8) | 30.6 (6.2)
Diabetes mellitus [Count of Participants; unit: Participants] | 18 | 15 | 33
Ejection fraction [Mean (Standard Deviation); unit: Percentage of blood] — Percentage of blood in the heart that is ejected out to the body with each heartbeat
  Percentage of blood | 57.8 (9.2) | 58.2 (9.6) | 58.0 (9.3)
MacNew Heart Disease Health-related Quality of Life questionnaire [Mean (Standard Deviation); unit: Units on a scale (7 point scale)] — A maximum score of 7 is associated with higher health related quality of life A minimum score of 1 is associated with poorer health related quality of life
  Units on a scale (7 point scale) | 2.7 (1.0) | 2.5 (0.8) | 2.6 (1.2)
Hypertension [Count of Participants; unit: Participants] | 44 | 43 | 87
Hyperlipidemia [Count of Participants; unit: Participants] | 45 | 40 | 85
Previous cardiac catheterization [Median (Inter-Quartile Range); unit: Days] | 37 [16 to 232] | 35 [23 to 73] | 36 [22 to 149]
Previous cardiac catheterization within 90 days preceding enrollment [Count of Participants; unit: Participants] | 40 | 38 | 78
Smoking [Count of Participants; unit: Participants]
  Past smoker | 28 | 19 | 47
  Active smoker | 6 | 3 | 9
Valvular heart disease [Count of Participants; unit: Participants] | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Steps
Description: The primary outcome variable is the change in mean daily step count from the baseline period to the maintenance period (weeks 9-16).
Time Frame: Baseline and end of Maintenance Period at Week 16
Measure: Mean (95% Confidence Interval); unit: Steps
Arm/Group | Control | Intervention
Number analyzed (Participants) | 55 | 50
Steps | 264 [95 to 433] | 1501 [1280 to 1722]

2. Secondary Outcome: Change in Mean Daily Steps From Baseline to Follow-up Period
Description: Secondary outcomes include change in mean daily steps from the baseline period to the follow-up period (weeks 17-24).
Time Frame: Baseline and end of Follow Up Period at week 24
Measure: Mean (95% Confidence Interval); unit: Steps
Arm/Group | Control | Intervention
Number analyzed (Participants) | 55 | 50
Steps | 92 [-236 to 420] | 1066 [885 to 1247]

ADVERSE EVENTS:
Time Frame: Through study completion (6 months).
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/50
Other Adverse Events (participants affected / at risk) | 0/55 | 0/50

LIMITATIONS AND CAVEATS:
Patients were from 4 hospitals in Southeastern Pennsylvania and had to use a smartphone or tablet. Physical activity measures were limited to only step counts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT02531022/Prot_SAP_000.pdf